CLINICAL TRIAL: NCT07130942
Title: The Effect of Inhalation Using a Molecular Hydrogen Generator on the Level of Exercise Capacity and Inflammatory Response, Anti-cancer Potential of Human Blood Serum in the Light of in Vivo/in Vitro Studies
Brief Title: Molecular Hydrogen Inhalation: Effects on Health, Exercise Capacity and Inflammatory Response - in Vivo/in Vitro Studies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: Medical University of Gdansk (Other); Kazimierz Wielki University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AWFiS/2025_8_JM
Record Dates: First submitted 2025-08-06; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Physiological Adaptations; Sport Performance; Aerobic Capacity; Anaerobic Power; Sport Recovery
Keywords: molecular hydrogen; anti-cancer potential; inflammatory response; exercise capacity; inhalation
MeSH Terms: conditions — Respiratory Aspiration | interventions — Hydrogen; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1-time molecular hydrogen inhalation intervention_SHAM intervention (Sham Comparator): 1 time SHAM intervention
  Interventions: Procedure: Inhalation using a molecular hydrogen generator
- Two weeks molecular hydrogen inhalation intervention_SHAM intervention (Sham Comparator): 14-days molecular hydrogen inhalation intervention
  Interventions: Procedure: Inhalation using a molecular hydrogen generator
- 1-time molecular hydrogen inhalation intervention (Experimental): 1-time molecular hydrogen inhalation intervention
  Interventions: Procedure: Inhalation using a molecular hydrogen generator
- Two weeks molecular hydrogen inhalation intervention (Experimental): 14-days molecular hydrogen inhalation intervention
  Interventions: Procedure: Inhalation using a molecular hydrogen generator

INTERVENTIONS:
Procedure: Inhalation using a molecular hydrogen generator — Hydrogen inhalation will be performed by using a hydrogen gas generator similar in terms of capabilities to the generator Hycellvator ET100 (Helix Japan, Co., Ltd., Tokyo, Japan). The apparatus will be generating 30.0 mL/s gas mixture, consisting of 68.0% hydrogen (hydrogen purity, 99.99%) and 32.0% of oxygen. All gases will be supplied through a nasal cannula connected to the gas generators. Although we could not measure directly the hydrogen and oxygen An average inspiratory flow rate will be adjusted to 500 mL/s at rest, the hydrogen concentration in the inspired gas must have been around 4.08% at most.
  Control population will have inhalation with the use of gas generator that has the same outer shape as the used generator to produce Placebo (30.0 mL/s, ambient air 400 m above sea level) consisting of 0.00005% of hydrogen and 20.9% of oxygen.
  Other Names: molecular hydrogen inhalation; molecular hydrogen therapy; Molecular hydrogen (H2) therapy

SUMMARY:
Summary To comprehensively address the research aims and explore the state of knowledge of the mechanisms of biochemical response to specific tissue affecting method in form of a molecular hydrogen inhalation and will allow to determine its role on the post-exercise response in form of changes in biochemical markers secretion, expression of selected trophic factors and changes in iron metabolism in this process.

Moreover, this project will try to take into account the role of hepcidin, vitamin D and cfDNA. Additionally, the present project may contribute to the determination of the role of presented inhalation procedure on cells proliferation, as example of anty-tumor proprieties, regulation of the expression of genes related to the stress response (HSF-1, NF-kB, TNF-dependent pathway), muscle cell growth (e.g. myostatin gene), energy pathways (e.g. GAPDH, LDH) and the membrane transport and the hedgehog pathway ls (including Gli1), Hif-1-alpha and NF-kB.

1.1. Primary Objectives

1. Demonstration relationship between post-exercise oxidative stress parameters, and two weeks of daily inhalation with the use of a molecular hydrogen generator.
2. Indicate of whether and how daily inhalation with the use of a molecular hydrogen generator will affect BDNF and hepcidin, erytropheron (ERFE) and erythropoietin (EPO).
3. Show how daily inhalation with the use of a molecular hydrogen generator and physical activity procedures effects human serum anti-tumor potential, and is it associated with Vitamin D status and Iron metabolism.

1.2. Secondary Objectives

1. Examine the relationship between two weeks of daily inhalation using a molecular hydrogen generator and the expression of genes related to the stress response (HSF-1, NF-kB, TNF-dependent pathway).
2. Show the relationship between the expression of genes related to muscle cell growth (e.g. myostatin gene), intracellular metabolism, energy pathways (e.g. GAPDH, LDH) and the effect of molecular hydrogen inhalation?
3. Show the molecular hydrogen inhalation effects on the expression of genes responsible for membrane transport and the hedgehog pathway in muscle cells (including Gli1), expression of transcription factors: Hif-1-alpha (hypoxia-inducible factor) and NF-kB and selected genes dependent on their activity.

1.3. Hypotheses

In the project on the basis of current knowledge, the following hypotheses are stated:

1. Daily inhalation with the use of a molecular hydrogen will increase the concentration of BDNF, which will correlate with higher skeletal muscle resistance to damage;
2. Two week daily inhalation with the molecular hydrogen will increase the concentration of BDNF, which will persist over a longer period compering to a single inhalation with the molecular hydrogen session;
3. Daily inhalation with the molecular hydrogen and physical activity effects on vitamin D binding protein, megalin, cubilin concentration changes.
4. Daily inhalation with the molecular hydrogen protects muscles and reduces oxidative stress induced by physical exercise and protects against oxidative stress induced by high Iron concentration (lower inflammation process and cfDNA concentration).
5. Daily inhalation with the molecular hydrogen effects human serum anti-tumor potential against human LNCaP prostate cancer cells.

III. Research project methodology In order to achieve the objectives of the study 80 people will be recruited, then randomly divided into two groups: Experimental ((N=40) and Control (N=40). Furthermore, groups will be divided into subgroups to implement the assumptions of one-time and 10-time inhalation with the use of a molecular hydrogen generator on the level of induced muscle damage and the level of maximum anaerobic and aerobic capacity. The whole study will be carried out using the assumptions of the experiment - a blind test (inhalation with normal air but under the use of H2 generator (switched of), and in accordance with the principles of the experiment.

In the study an experiment based on an ex post facto research plan will be used, due to the lack of manipulation of the grouping variable. Study will be based on comparative analysis and regression analysis. In the independent variable test, the group (non-trainees), variables dependent on molecular hydrogen inhalation and the anaerobic/aerobic performance characteristics, biochemical blood indicators. Minimal (40 people each) sample size was calculated according to Kirby et all (2002) and Kadam and Bhalerao (2010).

IV. The study will consist of twelve parts. For anaerobic power of the lower limbs measurement of double Wingate anaerobic test (WAnT) will be conducted on a cycle ergometer,

* For the measurement of Aerobic Components of Fitness and post-aerobic exercises response Bruce Treadmill Test will be performed.
* The blood collection for diagnostic tests will be strictly dependent on the requirements of a particular designation,

DETAILED DESCRIPTION:
1. RESEARCH PROJECT OBJECTIVES 1.1. Research project objectives The main aim of the project is to comprehensively evaluate the impact of molecular hydrogen inhalation on exercise capacity, inflammatory response, anti-tumour potential of human blood serum, and related molecular-genetic mechanisms involving oxidative stress, iron metabolism, gene expression regulation, and intracellular signalling pathways, assessed through in vivo and in vitro analyses.

The project aims to:

1. Demonstration relationship between oxidative stress parameters, uric acid concentration and nitric oxide degradation products in groups of people subjected to two weeks of daily inhalation with the use of a molecular hydrogen generator.
2. Indicate of whether and how one time and daily inhalation with the use of a molecular hydrogen generator will affect BDNF and hepcidin concentration, and whether these changes will be accompanied by greater resistance of skeletal muscles to damage induced by exercises;
3. Show whether two weeks daily inhalation with the use of a molecular hydrogen generator will induce a higher changes of BDNF, hepcidin erytropheron (ERFE) and erythropoietin (EPO) concentration (compared to a single session of inhalation with the use of a molecular hydrogen);
4. Show how daily inhalation with the use of a molecular hydrogen generator and physical activity procedures effects human serum anti-tumour potential, and is it associated with Vitamin D status and Iron metabolism.
5. Show is there a relationship between one time and two weeks of daily inhalation using a molecular hydrogen generator and the expression of genes related to the stress response (HSF-1, NF-kB, TNF-dependent pathway).
6. Show the relationship between the expression of genes related to muscle cell growth (e.g. myostatin gene) and the effect of molecular hydrogen inhalation?
7. Demonstrate the relationship between the expression of genes related to intracellular metabolism and the effect of molecular hydrogen inhalation.
8. Show the relationship between the expression of genes encoding enzymes of energy pathways (e.g. GAPDH, LDH) and the effect of molecular hydrogen inhalation in the study group
9. Show the molecular hydrogen inhalation effects on the expression of genes responsible for membrane transport and the hedgehog pathway in muscle cells (including Gli1), expression of transcription factors: Hif-1-alpha (hypoxia-inducible factor) and NF-kB and selected genes dependent on their activity.

1.2. Hypotheses

In the project on the basis of current knowledge, the following hypotheses are stated:

1. Daily inhalation with the use of a molecular hydrogen will increase the concentration of BDNF, which will correlate with higher skeletal muscle resistance to damage;
2. Two week daily inhalation with the molecular hydrogen will increase the concentration of BDNF, which will persist over a longer period compering to a single inhalation with the molecular hydrogen session;
3. Daily inhalation with the molecular hydrogen and physical activity effects on vitamin D binding protein, megalin, cubilin concentration changes.
4. Daily inhalation with the molecular hydrogen protects muscles and reduces oxidative stress induced by physical exercise and protects against oxidative stress induced by high Iron concentration (lower inflammation process and cfDNA concentration).
5. Daily inhalation with the molecular hydrogen effects human serum anti-tumor potential against human LNCaP prostate cancer cells.

2. SIGNIFICANCE OF THE PROJECT Physical performance, encompassing endurance, muscle strength, and explosive power, serves as a fundamental element for success in sports among both non-athletic individuals and athletes.

It not only enhances competitive performance on the field but also encourages healthy adults to engage in sports. Oxidative stress arises when the products of oxygen metabolism accumulate and exceed the body's ability to resist oxidation. Research indicates that physical activity at varying intensities can influence the levels of different oxidative biomarkers.

Nevertheless, engaging in physical exercise, particularly at moderate to high intensities, may result in excessive oxidative stress, adversely affecting redox homoeostasis, increasing fatigue, and ultimately diminishing physical performance.

Consequently, there has been a focus on investigating potential antioxidant strategies to develop effective methods for improving physical performance. Molecular hydrogen (H2) has emerged as a promising antioxidant that selectively neutralises hydroxyl radicals and peroxynitrite in cells without diminishing other reactive species.

The suggested benefits of molecular hydrogen in the body, are due the fact that H2 is a potent antioxidant and signalling molecule. Unlike conventional antioxidants that non-selectively scavenge reactive oxygen species (ROS) and reactive nitrogen species (RNS), hydrogen selectively targets highly reactive and deleterious species such as hydroxyl radicals (•OH) and peroxynitrite (ONOO-), thereby preserving ROS involved in physiological signalling, which is crucial for cellular homoeostasis and adaptation. Recent studies have shown that modulating ROS and subsequently regulating the gas transmitters nitric oxide and carbon monoxide to influence NO-CO metabolism may have beneficial effects on various diseases. Studies have shown that molecular hydrogen, which can be delivered to the body in various forms (i.e. inhaled gas - H2 inhalation, drinking hydrogen-rich water (HRW) and intravenously in H2 saline solution), can penetrate cell membranes and rapidly diffuse into cellular organelles (e.g. mitochondria), thereby increasing the functional efficiency of mitochondria and enhancing ATP production or lactate oxidation. Recent human studies have begun to investigate the potential advantages of H2 for enhancing physical performance, showing significant promise for H2-based interventions. However, the findings and study designs regarding the impact of H2 on physical performance have varied.

Regulation of gene expression: ROS play a role in the regulation of gene expression, particularly in genes involved in stress responses and antioxidant production. By maintaining physiological levels of ROS, hydrogen can aid in the proper regulation of these genes, supporting cellular defence mechanisms and resilience against oxidative stress. Overall, these beneficial properties not only protect cells from oxidative damage but also support critical signalling pathways that promote health, adaptation, and recovery.

The potential effects of molecular hydrogen on exercise physiology are multifaceted, influencing a wide range of physiological processes encompassing energy metabolism, oxidative stress modulation, inflammation regulation, cell signalling modulation, and recovery facilitation mechanisms. By regulating these key pathways, molecular hydrogen offers an alternative approach to optimising athletic performance, mitigating exercise-induced muscle damage and accelerating post-exercise recovery.

Despite growing interest in this area, several fundamental questions remain unanswered]. A primary concern is determining which specific exercise patterns-aerobic, anaerobic derive the most benefit from molecular hydrogen inhalation. It is well established that sports encompass a diverse range of activities, each requiring distinct skills such as cardio respiratory fitness, muscular strength, muscular endurance, flexibility, agility, coordination, power, reaction time, and speed. However, the extent to which HRW can enhance these specific skills remains unclear and warrants further investigation. Additionally, to effectively develop of molecular hydrogen inhalation procedure as improving sport result procedure and promote its use among a broader athletic audience, it is crucial to identify the specific physiological advantages that might enhance athletic performance.

Recent years brought the era of cell-free DNA (cfDNA) as a potential biomarker of the level of injury, which is gaining interest in many various biomedical disciplines, including the field of exercise physiology. There are more and more studies looking for the role of cfDNA as a potential hallmark of the overtraining syndrome in: resistance training, marathon run, continuous treadmill running, incremental exercise, rowing exercise, strength training.

Besides cfDNA might be related to, or trigger adaptations of immune function induced by strenuous exercise. Publication from 2017 revealed an increase cf-DNA level even during aerobic running below the lactate steady state depending on intensity and duration. It was observed that cfDNA concentrations peaked immediately after acute exercise and about 1h post-exercise returned to baseline levels. Furthermore, typical markers of skeletal muscle damage (C-reactive protein, uric acid, creatine kinase, myoglobin) display delayed kinetics compared with the cfDNA peak response. All of that underlines the potential of cfDNA as a biomarker for exercise load in both-the aerobic and the anaerobic state. However, there was not much effort put into finding the correlations between cf-DNA and iron state and exercises induced inflammation process.

This project will have an impact on the development of the current state of knowledge of the mechanisms of biochemical response to specific tissue affecting method in form of a molecular hydrogen inhalation and will allow to determine its role on the post-exercise response in form of changes in biochemical markers secretion, expression of selected trophic factors and changes in iron metabolism in this process. Moreover, this project will try to take into account the role of hepcidin, vitamin D and cfDNA. Additionally, the present project may contribute to the determination of the role of presented inhalation procedure on cells proliferation, as example of ant-tumour proprieties, regulation of the expression of genes related to the stress response (HSF-1, NF-kB, TNF-dependent pathway), muscle cell growth (e.g. myostatin gene), energy pathways (e.g. GAPDH, LDH) and the membrane transport and the hedgehog pathway ls (including Gli1), Hif-1-alpha and NF-kB.

Therefore, the results of this project could be a significant step in expanding our understanding of the role of molecular hydrogen inhalation in the healthy population (in modulating post-exercise muscle damage, cells proliferation, inflammation process) and the role of iron metabolism and vitamin D in those changes. In addition, the knowledge on the protective effect of molecular hydrogen inhalation procedures and their relation to BDNF changes and protein kinase activity will give us overview of its novel activity and use.

The research team involved in this project possesses extensive expertise and significant experience confirmed by numerous scientific publications, particularly in the field of human physiology, exercise-induced adaptive responses, and various intervention strategies aimed at optimising recovery and performance. Members of the team have previously published research on oxidative stress modulation, inflammatory responses, genetic expression changes, and biochemical adaptations following physical exercise, ensuring that the methodologies and analytical approaches proposed in this study are robust, reliable, and scientifically validated

3. WORK PLAN In order to achieve the objectives of the study the minimal population sample size allowing to support the appropriate power of the study of interactions between the effects was calculated using GPower ver. 3.1.9.2 software. The minimal sample size was 64 people. Due to the possibility of participants not completing the project, a 20% population increase was assumed in order to obtain the desired study size population of 80 people will be recruited, then randomly divided into two groups: Experimental (N=40) and Control (N=40).

Furthermore, groups will be divided into subgroups to implement the assumptions of one-time and 10-time inhalation with the use of a molecular hydrogen generator on the level of a induced muscle damage and the level of maximum anaerobic and aerobic capacity. The whole study will be carried out using the assumptions of the experiment - a blank test, and in accordance with the principles of the cross-fertilisation experiment.

3.1 Compliance and Monitoring: To ensure adherence to protocols and maintain the integrity of the study, compliance will be carefully monitored through various measures. Weekly participant check-ins will be conducted to track progress and confirm adherence to the study protocols. Digital logs will document exercise routines and dietary compliance, providing a transparent record of participant engagement throughout the study period. Real-time monitoring during supervised sessions will verify the accurate implementation of exercise and inhalation procedures. In the case of participant dropouts, replacements will be identified through re-screening to preserve statistical validity and ensure that the required sample size is maintained. Additionally, a clinical and sports dietitian will continuously assess dietary adherence and make necessary adjustments to the dietary plans, ensuring consistency and compliance across the study population.

3.2. Experiment Plan:

1. Enrolment of the participants - All untrained subjects will be selected on the basis of the intent letter.
2. Laboratory measurements

   1. anaerobic test (Wingate Anaerobic Test), 1 time H2 inhalation, two-weeks H2 inhalation, anaerobic test (Wingate Anaerobic Test),
   2. aerobic test (Bruce Aerobic test), 1 time H2 inhalation, two-weeks H2 inhalation, anaerobic test
   3. evaluation of human serum (from one-time, two-weeks H2 inhalation and placebo populations) anti-tumour potential on human LNCaP prostate cancer cells
3. Blood chemistry and molecular analysis
4. Analysis and interpretation of results, preparation of scientific publications 5. Preparation of scientific publications, project settlement.

   3.3 Risk Management Plan for the research project 3.3.1. Risk Identification • Technical risk: laboratory equipment failures, software problems, calibration problems, incorrect data processing.
   * Risks related to research on humans: The project includes potential physical and psychological risks, mainly related to intense physical exercise. Moreover, there is a risk of the participant not completing the research.
   * Financial risks: budget overruns, insufficient funds.
   * Schedule risks: delays in the implementation of tasks, problems with the availability of the research entity, problems with the availability of services related to the implementation of the project: medical services, services related to the indicated measuring devices.
   * Organization all risks: changes in the project team, communication problems,
   * External risks: changes in legal regulations, unfavourable weather conditions, market changes.

   3.3.2. Prevention and Corrective Actions

   Hardware failures:
   * Prevention: Regular inspections and maintenance of equipment, having spare devices, scientific partnership with the Medical University of Gdańsk, Laboratory of Physical Exercise and Genetics in Sports of the Gdansk University of Physical Education and Sport in Gdańsk - has current equipment inspections, contracts.
   * Correction: Quick repair or replacement of damaged equipment within 14 days, contract with an external service (Institutional agreements).

   Risks associated with research on humans:

   • Prevention: All procedures will be carried out in accordance with the approved protocol by the Bioethics Committee. Participants will be thoroughly informed about the procedures, potential risks and benefits before giving informed consent. Presence of qualified medical personnel during stress tests. According with the statistical calculations necessary population (number of participants needed to achieve statistical significance) for the research is much lower that the prospective recruited.

   • Correction: Participants will be monitored throughout the study (both by the experimental teem and study assistance and medical attention will be provided as needed. During all stages of the experiment all participants will be provided with care to ensure their comfortable participation and to solve any problems that may arise during experiment.

   Risks associated with intense physical exercise
   * Intense exercise, both anaerobic and aerobic, can lead to injuries, overuse and other health problems such as heart rhythm disturbances, excessive fatigue or dehydration and many other.
   * Prevention: Conducting preliminary medical examinations by professional medical doctor (to exclude participants with contraindications to intense physical exercise). Constant monitoring of participants' vital parameters during tests, medical care at every stage of research experiments .
   * Correction: Immediate medical intervention if symptoms of excessive fatigue or injury occur Risk associated with blood collection for the purpose of separating blood serum
   * Blood collection is a procedure related to disruption of skin and tissue continuity, which may cause pain, bleeding and other complications (including bruising, soreness, etc.).
   * Prevention: Blood collection performed by experienced specialists in sterile conditions. Close monitoring of the blood collection site during the collection period and the time interval after collection.
   * Correction: Immediate medical intervention-related complications (compression, elevation, cooling, use of dressings that accelerate blood clotting).

   Risk related to the participant's failure to complete the research due to unforeseen circumstances
   * Prevention: Recruiting more participants than the required minimum study sample to minimise the impact of participant dropouts or exclusions on study results. Conducting thorough screening of participants based on their health status, medical history, motivation and availability to minimise the risk of non-completion of the study. Providing participants with regular psychological and motivational support throughout the duration of the study.
   * Correction: If a participant drops out or is excluded at the beginning of the study, replace him or her with a new participant who meets the study criteria. If necessary, flexible adjustment of the study schedule for participants who have difficulty meeting deadlines.

   Overspend:
   * Prevention: Careful cost analysis before project initiation and regular monitoring of expenses within available supplies of reagents and consumables.
   * Correction: Searching for additional sources of financing, negotiations with suppliers as part of the pricing policy, searching for alternative marking methods of similar quality but less costly.

   Delays in the implementation of tasks:

   • Prevention: Realistic planning of the testing schedule, ensuring qualified medical personnel during exercise tests and tissue collection. In case of absence, providing possible replacements.

   • Correction: Assigning additional human resources to critical tasks. 3.4. Milestones of the study

   • Project approval by Bioethics Committee (achieved before starting the project - a necessary condition for carrying out the study; Bioethics Committee);

   • Recruitment for research (the initial recruitment carried out allows the effectiveness of targeted recruitment to the study to be highly probable; all study procedures are well known for the researchers and won't create any problems - ); during the initial recruitment for the project, 80 people were recruited to actively participate in the study;

   • Funding (achieving funding will allow us to proceed with the research);

   • Assessment of the maximum anaerobic and aerobic capacity (research procedures carried out during the study do not differ from other generally accepted studies carried out by members of the research team, allowing for the assumption of full success in the implementation of the study)

   • Evaluation of selected biochemical samples ( the proposed research methods in the implemented protocol are characterised by high selectivity and high research quality, allowing the obtaining valuable scientific results)

   • Finalisation of the project's research tasks (the obtained results allow the acceptance or rejection of the proposed research hypotheses regardless of the nature of the observed changes) 3.5. Deliverables of the study

   • Tangible deliverables: full blood samples, serum samples, cfDNA samples, obtained results from immunoenzymatic, mass spectroscopic and biochemical analyses, results from maximal anaerobic and aerobic testing, research results and conclusions from them, written publications, practical guidelines for performing the exercises
   * Intangible deliverables: new knowledge and practical skills, of the research team members, knowledge of the participants in the research project about the inhalation procedures that can be performed in home conditions.

   3.5 Project management Use the critical path method to highlight all of the tasks that are absolutely necessary for the project's completion (according to the research plan and research task). This type of project management will help the whole research team to identify the most optimal workflow to create an efficient project timeline (according to the plan).

   According to the project management, critical path tasks are:
   * recruitment of study populations and its randomisation (with the resource buffers);
   * performance of exercises testing and sample collection (validated testing methods that were performed previously),
   * securing research samples (resource buffers - 4 copies of every sample in different fringes);
   * recruitment of study populations and its randomisation (with the resource buffers);
   * performance of exercises testing and sample collection (validated testing methods that were performed previously),
   * analyses of the samples (use only the analytical methods with high-quality results and repeatability of measurements);
   * statistical analysis based on consultation with a bio-statisticia,
   * discussion of the obtained results during a discussion panel of all researchers implementing the research to maintain high quality and reliability of results and conclusions)
   * preparation of publications and their submission to journals of high scientific level.

4. RESEARCH METHODOLOGY In the study an experiment based on an ex post facto research plan will be used, due to the lack of manipulation of the grouping variable. Study will be based on comparative analysis and regression analysis. In the independent variable test, the group (non-trainees), variables dependent on molecular hydrogen inhalation and the anaerobic/aerobic performance characteristics, biochemical blood indicators.

In order to implement the assumptions of the study, min. 80 people will be recruited, randomly divided into two groups, a minimum of 40 people in each:

* EXPERIMENTAL (E1; E10)- single session of a molecular hydrogen inhalation and two-week daily inhalation with the use of a molecular hydrogen generator (N=40),
* CONTROL GROUP (C1; C10) (N=40),

The whole study will be carried out using the assumptions of the experiment - a blind test (inhalation with normal air but under the use of H2 generator (switched of), and in accordance with the principles of the experiment.

4.1 Material INCLUSION CRITERIA - PHYSICAL ACTIVE, NOT TRAINING GROUP

The study will be used purposeful selection of the following criteria:

* age 18-25,
* not taking medicines during the study,
* negative history of cardiovascular disorders,
* negative history of autonomic nervous system disorders,
* negative history of mental disorders,
* negative history of cerebra-cranial traumas,
* negative history of other diseases that may directly affect obtained results,
* good health status (no concurrent injuries);'
* no drugs intake,
* no supplements consumption,

In the study as a not training grope age and morphologically appropriate participation will take part. Participants will be recruited basing on a voluntary letter of intent. All representatives of the analysed group participating in the pre-qualification research will fill in the physical activity sheet - Global Health Activity Questionnaire - World Health Organization in Polish adaptation. This will allow to eliminate people who report high levels of physical activity (similar to the level of sport training individuals).

4.2. Procedures

The study will consist of twelve parts:

1. assessment of general health (medical examination), and familiarisation with detailed study protocol;
2. assessment of the maximum anaerobic capacity (WAnT);
3. assessment of one-time and two-weeks of molecular hydrogen inhalation;
4. evaluation of the impact of one time and two-weeks of molecular hydrogen inhalation procedure on WAnT testing, the level of inflammatory response markers, iron homoeostasis, vit D metabolites, BDNF, selected genes expression in research in selected time points tested.
5. evaluation of human serum (from one time and two-weeks of molecular hydrogen inhalation and placebo populations) anti-tumour potential on human LNCaP prostate cancer cells;
6. evaluation of selected laboratory exponents in serum and plasma samples collected during the study 24 hours, 48 hours, 72 hours and 120 hours from an episode of muscle damage induced by eccentric exercises; Two-months pause

<!-- -->

1. assessment of general health (medical examination), and familiarisation with detailed study protocol;
2. assessment of the maximum aerobic capacity (Bruce test);
3. assessment of one-time and two-weeks of molecular hydrogen inhalation
4. evaluation of the impact of one time and two-weeks of molecular hydrogen inhalation procedure on WAnT testing, the level of inflammatory response markers, iron homoeostasis, vit D metabolites, BDNF, selected genes expression in research in selected time points tested.
5. evaluation of human serum (from one time and two-weeks of molecular hydrogen inhalation and placebo populations) anti-tumor potential on human LNCaP prostate cancer cells;
6. evaluation of selected laboratory exponents in serum and plasma samples collected during the study 24 hours, 48 hours, 72 hours and 120 hours from an episode of muscle damage induced by eccentric exercises; Each participant will be at hydrated state and before their first meal in the morning hours. Before proper measures, each participants had one week earlier a familiarisation session with all procedures.

   4.3. Molecular hydrogen inhalation procedures. Hydrogen inhalation will be performed by using a hydrogen gas generator similar in terms of capabilities to the generator Hycellvator ET100 (Helix Japan, Co., Ltd., Tokyo, Japan). The apparatus will be generating 30.0 mL/s gas mixture, consisting of 68.0% hydrogen (hydrogen purity, 99.99%) and 32.0% of oxygen. All gases will be supplied through a nasal cannula connected to the gas generators. Although we could not measure directly the hydrogen and oxygen An average inspiratory flow rate will be adjusted to 500 mL/s at rest, the hydrogen concentration in the inspired gas must have been around 4.08% at most.

   Control population will have inhalation with the use of gas generator that has the same outer shape as the used generator to produce Placebo (30.0 mL/s, ambient air 400 m above sea level) consisting of 0.00005% of hydrogen and 20.9% of oxygen.

   4.4. Measurement of anaerobic power of the lower limbs For anaerobic power of the lower limbs measurement of double Wingate anaerobic test (WAnT) will be conducted on a cycle ergometer. Before any experimental testing, each individual will perform a 5 min warm-up on the cycle ergometer with tempo of 60 rpm and 1W/kg. After five minutes break, each participant will be asked to pedal with maximum effort for a period of 30 s against a fixed resistive load of 75 g/kg of total body mass. After finishing the test 30 s pause will began and second WAnT performance will be made.

   Each participant was instructed to cycle as fast as possible and was given a 3s countdown before the set resistance was applied Verbal encouragement will be given to all participants to maintain their highest possible cadence throughout WAnT. Data from the cyclo-ergometer will be recorded via computer with the MCE 5.1 software.

   The following WAnT variables will be considered:

   • total work value (Wtot),

   • maximum anaerobic power (PPWAnT),

   • maximum power (TUZ),

   • maximum power maintenance (TUT) to 0.01s,
   * power drop (WSM) (%). Variables will be analysed as absolute values (W) and relative to body mass (W/kg).

   4.5 Measurement of of Aerobic Components of Fitness For the measurement of Aerobic Components of Fitness and post-aerobic exercises response Bruce Treadmill Test will be performed. The Bruce protocol will be performed on an electric treadmill (H/P/Cosmos, München, Germany) one months after WAnT procedure.

   4.6 Blood samples collection and measurements The methodology of blood collection for diagnostic tests will be strictly dependent on the requirements of a particular designation and comply with the research procedures (established on the basis of literature data). For laboratory analysis, peripheral blood will be collected. in accordance with the plan. Aerobic and anaerobic components of fitness will be tested with two month will be tested with a 2 month break between each testing and inhalation with H2 • for WAnT: before physical exercise, immediately after completion of the Wingate test (up to 5 minutes after the test), after 30 minutes of rest period after completion of the Wingate test (30-35 minutes after the test), 60 minutes after, 6h after, 24 hours after WAnT, • for Bruce Treadmill Test: before physical exercise, immediately after completion of the Bruce trial (up to 5 minutes after the test), after 30 minutes of rest period after completion of the test (30-35 minutes after the test), 60 minutes after, 6h after, 24 hours after the trial,

   The intake will be performed in appropriate standardised BD Vacutainer tubes by qualified medical personnel.

   Serum and plasma will be separated from the samples, Each sample to obtain the serum will be centrifuged at 2500-3000 rpm for 10 minutes in 4° C and stored in Eppendorf tubes at - 80° C until the assay (no longer than 6 months).

   The following secretory factors and markers of inflammation will be determined in serum or blood plasma (depending on the requirements of the method used) and then analysed in detail:

   • hsCRP, CK, lactic acid, IL-6, IL-10, TNF-α, Irisine, BDNF,
   * hepcidin, TIBC, transferrin, ferritin, EPO, EFRE,
   * vit D binding protein, 25(OH)D3, 24,25(OH)2D3, 3-epi-25(OH)D3, and 25(OH)D2 levels; and the ratios of 25(OH)D3 to 24,25(OH)2D3, and 25(OH)D3 to 3-epi-25(OH)D3

   The general assessment of the homoeostasis state will be based on preliminary laboratory tests such as:

   • blood morphology, glycaemic, activity of ALT, AST, CK, LDH, concentration of insulin, total cholesterol, creatine.

   For the qualitative detection of single proteins involved in antioxidant defence western blotting technique will be performed. Proteins involved in antioxidant defense, and inflammation will be identified and measured.
   * involved in antioxidant defense (SOD1, SOD2, GPx),
   * inflammation (IL-6). cfDNA will be collected into cell-free DNA tubes and isolated using Quick-cfDNA Serum & Plasma Kit according to the manufacturer's protocol.

   4.8. Cytotoxic activity The cytotoxic activity will be evaluated using the method described by Paredes-Gamero et al.

   4.9 Statistical analysis The results will be analysed statistically using Statistica software. Statistical significance will be determined for p < 0.05. The project analyses significance of differences in results, WAnT and laboratory parameters between groups; Significance of changes after WAnT and regression analysis of test results.

ELIGIBILITY:
Inclusion Criteria:

The study will be used purposeful selection of the following criteria:

* age 18-25,
* not taking medicines during the study,
* negative history of cardiovascular disorders,
* negative history of autonomic nervous system disorders,
* negative history of mental disorders,
* negative history of cerebrospinal traumas,
* negative history of other diseases that may directly affect obtained results,
* good health status (no concurrent injuries),
* no drugs intake,
* no supplements consumption,

In the study as a not training grope age and morphologically appropriate participation will take part. Participants will be recruited basing on a voluntary letter of intent. All representatives of the analysed group participating in the pre-qualification research will fill in the physical activity sheet - Global Health Activity Questionnaire - World Health Organization in Polish adaptation. This will allow to eliminate people who report high levels of physical activity (similar to the level of sport training individuals).

Exclusion Criteria:

* taking medicines during the study,
* history of cardiovascular disorders,
* history of autonomic nervous system disorders,
* history of mental disorders,
* history of cerebrospinal traumas,
* history of other diseases that may directly affect obtained results,
* concurrent injuries,
* drugs intake,
* supplements consumption.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-09-28 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of the inflammation blood markers using Magnetic Luminex Performance Assays | Change from baseline at 24 hours after fatigue-induced exercise (before and after each protocol)
  The intake will be performed in appropriate standardized BD Vacutainer tubes by qualified medical personnel: Serum and plasma will be separated from the samples, Each sample to obtain the serum will be centrifuged at 2500-3000 rpm for 10 minutes in 4° C and stored in 1.5 ml tubes at - 80° C until the assay (no longer than 6 months). The following secretory factors and markers of inflammation will be determined in serum or blood plasma (depending on the requirements of the method used) and then analysed in detail using immu: • high sensitive C-protein (hsCRP), • creatine kinas (CK), • lactic acid (LA), • interleukin 6 (IL6), • interleukin 10 (IL10), • interleukin 15 (IL15),
Measurement of the Iron metabolism blood markers using Magnetic Luminex Performance Assays and ELISA Assays | Change from baseline at 24 hours after fatigue-induced exercise (before and after each protocol)
  The intake will be performed in appropriate standardized BD Vacutainer tubes by qualified medical personnel: Serum and plasma will be separated from the samples, Each sample to obtain the serum will be centrifuged at 2500-3000 rpm for 10 minutes in 4° C and stored in 1.5 ml tubes at - 80° C until the assay (no longer than 6 months). The following secretory factors and markers will be messured: • free Iron • hepcidin, • transferrin, • ferritin, • EPO, • EFRE, • TIBC,
Measurement of neurotrophic, angiogenic blood markers using Automated Hematology Analyzers and Magnetic Luminex Performance Assays | Change from baseline at 24 hours after fatigue-induced exercise (before and after each protocol)
  The intake will be performed in appropriate standardized BD Vacutainer tubes by qualified medical personnel: Serum and plasma will be separated from the samples, Each sample to obtain the serum will be centrifuged at 2500-3000 rpm for 10 minutes in 4° C and stored in 1.5 ml tubes at - 80° C until the assay (no longer than 6 months). The following secretory factors and markers of inflammation will be determined: angiogenin (ANG), • insulin-like growth factor-1 (IGF-1), • Growth Differentiation Factor 15 (GDF15), • nerve growth factor (NGF), • Amyloid Precursor Protein- α (sAPPα), • angiopoietin (ANGP1), • brain-derived neurotrophic factor (BDNF) • growth differentiation factor 15 (GDF-15), • tumor necrosis factor α (TNFα).
The general assessment of the homoeostasis Automated Hematology Analyzers | Before all procedures and before post-hydrogen inhalation testing
  • blood morphology, • glycemia, • free iron, • activity of alanine aminotransferase (ALT), • aspartate aminotransferase (AST), • creatine kinase (CK), • lactate dehydrogenase (LDH), • concentration of insulin, • total cholesterole • creatinine,

SECONDARY OUTCOMES:
Measurement of proteins involved in antioxidant defence using Western Blotting Techniques | Before and after 1-time and 14-times inhalation using a molecular hydrogen generator
  Description: Qualitative detection of single proteins involved in antioxidant defence using western blotting technique. Proteins involved in antioxidant defence, and inflammation will be identified and measured: • involved in antioxidant defense (superoxide dismutase [SOD1], SOD2, glutathione peroxidase [GPx]), • inflammation (interleukin-6).
Messurment of cfDNA changes | Before, and 5 min, 60 min after every WAnT and Bruce Test performance
  cfDNA will be collected into cell-free DNA tubes (Roche) and isolated using Quick-cfDNA Serum & Plasma Kit (Zymo Research) according to the manufacturer's protocol. Obtained material will be aliquoted, stored in -200C and subsequently used for further analyses. Blood samples will be collected into cell-free DNA tubes before physical exercise (in the morning, on an empty stomach), immediately after the end of trial, 5 minutes and 60 minutes after the end of exercise. Collected material will be stored in a refrigerator or on ice for cfDNA isolation
Measurement of isolated serum cytotoxic activity | Up to 12 months post-experimental period
  The LNCaP cell line will be cultured in RPMI 1640 medium supplemented with 10% fetal bovine serum (FBS), 100 U/mL of penicillin, and 100 μg/mL of streptomycin, and incubated in a humidified atmosphere at 37°C and 5% CO2. The cytotoxic activity will be evaluated using the method described by Paredes-Gamero with some modifications. Cells will be plated onto 96-well microplates (105 cells/mL) in RPMI 1640 supplemented with 10% FBS in the absence or presence of the EEHS (25-200 μg/mL) for 24 h in a humidified atmosphere at 37°C and 5% CO2. After this period, the cells will be washed with PBS and resuspended in buffer (0.01 M HEPES, pH = 7.4, 0.14 M NaCl and 2.5 mM CaCl2). The stained cells will be fluorescently labeled and analyzed using an Accuri C6 flow cytometer and Accuri C6 software.

OTHER OUTCOMES:
Body composition analyses using bioelectrical impedance analysis (BIA) | During the initial visit, and before and after every experimental phase (1-time; 14-times inhalation using a molecular hydrogen generator)
  The participant's body mass and height, leg lean mass (LLM) of lower limbs will be measured by a multi-frequency bioelectrical impedance method using the body composition analyser - Inbody 720 (Biospace, Korea, Seoul). Weight and height will be combined to report BMI in kg/m^2, and all specific analyses will give percent of muscle mass in every limb and part of body. The measured values will be served for normalisation of the peak torque outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jędrzej Antosiewicz, Full Profesor, Principal Investigator — Medical University of Gdańsk, Department of Bioenergetics and Physiology of Exercise, Gdańsk, Poland
Locations (1):
- University of Physical Education and Sport (GUPES), Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared only on rational wishes from the main researchers

REFERENCES:
- [Background] Chomczynski P, Sacchi N. Single-step method of RNA isolation by acid guanidinium thiocyanate-phenol-chloroform extraction. Anal Biochem. 1987 Apr;162(1):156-9. doi: 10.1006/abio.1987.9999. PMID 2440339
- [Background] Sim M, Kim CS, Shon WJ, Lee YK, Choi EY, Shin DM. Hydrogen-rich water reduces inflammatory responses and prevents apoptosis of peripheral blood cells in healthy adults: a randomized, double-blind, controlled trial. Sci Rep. 2020 Jul 22;10(1):12130. doi: 10.1038/s41598-020-68930-2. PMID 32699287
- [Background] Farley JB, Stein J, Keogh JWL, Woods CT, Milne N. The Relationship Between Physical Fitness Qualities and Sport-Specific Technical Skills in Female, Team-Based Ball Players: A Systematic Review. Sports Med Open. 2020 Apr 15;6(1):18. doi: 10.1186/s40798-020-00245-y. PMID 32297147
- [Background] Timon R, Olcina G, Gonzalez-Custodio A, Camacho-Cardenosa M, Camacho-Cardenosa A, Martinez Guardado I. Effects of 7-day intake of hydrogen-rich water on physical performance of trained and untrained subjects. Biol Sport. 2021 Jun;38(2):269-275. doi: 10.5114/biolsport.2020.98625. Epub 2020 Oct 22. PMID 34079172
- [Background] Botek M, Khanna D, Krejci J, Valenta M, McKune A, Sladeckova B, Klimesova I. Molecular Hydrogen Mitigates Performance Decrement during Repeated Sprints in Professional Soccer Players. Nutrients. 2022 Jan 25;14(3):508. doi: 10.3390/nu14030508. PMID 35276867
- [Background] Itoh T, Hamada N, Terazawa R, Ito M, Ohno K, Ichihara M, Nozawa Y, Ito M. Molecular hydrogen inhibits lipopolysaccharide/interferon gamma-induced nitric oxide production through modulation of signal transduction in macrophages. Biochem Biophys Res Commun. 2011 Jul 22;411(1):143-9. doi: 10.1016/j.bbrc.2011.06.116. Epub 2011 Jun 23. PMID 21723254
- [Background] Hancock JT, Russell G. Downstream Signalling from Molecular Hydrogen. Plants (Basel). 2021 Feb 14;10(2):367. doi: 10.3390/plants10020367. PMID 33672953